CLINICAL TRIAL: NCT06773169
Title: IAMABLE: Implementation and Evaluation of an App for Evidence-Based Self-Management Rehabilitation Strategies
Acronym: IAMABLE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PJT-195979; PJT-195979 (Other Grant/Funding Number: Canadian Institutes for Health Research)
Record Dates: First submitted 2025-01-06; First posted 2025-01-14 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Neurological Conditions; Musculoskeletal Diseases or Conditions; Cardiovascular Diseases
Keywords: rehabilitation; chronic conditions; self-management; technology; web-based application
MeSH Terms: conditions — Musculoskeletal Diseases; Cardiovascular Diseases; Chronic Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IAMABLE Group (Experimental): The IAMABLE Group will use the IAMABLE app to engage in self-management.
  Interventions: Other: IAMABLE web-based app
- Control Group (Sham Comparator): The Control Group will receive general health information.
  Interventions: Other: General health information

INTERVENTIONS:
Other: IAMABLE web-based app — The Intervention Group will use the IAMABLE app for 4 months. IAMABLE users identify activities that they are having difficulty with because of their health problem and set goals they want to work toward. Self-management (SM) modules help them reach their goals, providing information and rehabilitation strategies about exercise, fall prevention, fatigue management, pain management, physical activity, and stress management. Users complete a self-assessment associated with each module, and receive tailored recommendations that guide them to access relevant module topics. Users create 7-day action plans using the strategies in the module to address their activity goals. Users receive automated notifications when it is time to evaluate action plans and activity goals, as well as weekly messages to remind them to engage with the app. Users have access to therapist support using the Ask a Therapist feature and receive individual consultations in response to queries about SM.
  Arms: IAMABLE Group
Other: General health information — The Control Group will receive a monthly email with general health information (not specific to rehabilitation or chronic diseases) for 4 months. Topics will include Nutrition, Vision Care, Foot Care, Hearing, Skin Care and Oral Care. Each email will include an introduction to the topic and links for additional information.
  Arms: Control Group

SUMMARY:
Background: As the population gets older, a rise in chronic conditions has resulted in increased demand for rehabilitation. We developed a web-based app called IAMABLE (I am able), to share evidence-based rehabilitation strategies with people with chronic conditions. Our project will guide us to test this app's effectiveness and explore the ways that people use it.

Goals, Methods, Approach: This pilot randomized controlled trial will offer people receiving the intervention access and use of the IAMABLE app for 4 months. People in the comparison group will have access to general web-based health information. We will recruit 50 people, 45 to 75 years, with at least one chronic condition; we will advertise in five communities (Hamilton, Kingston, London, Halifax, Winnipeg) to evaluate feasibility of the study design.

Patients, therapists and app experts will be an expert group to study how the app encourages people to start and continue to use it. We will use patient-reported measures to determine if the people in the IAMABLE group experience better function; quality of life, mobility, participation, self management, pain, health service use, and falls are secondary outcomes. We will measure outcomes at baseline, 4 and 8 months.

Research Team: Our team is led by researchers with experience in rehabilitation and chronic disease management, including testing technology innovations. Patient advisors will support the project, along with co-investigators with expertise in statistics, technology, and rehabilitation research.

Expected Outcomes: This research has the potential to prove how a web-based app can deliver occupational therapy and physiotherapy to support health and well being for people with chronic conditions. After this study, we plan a larger trial that will focus on effectiveness and address sustained use. IAMABLE will become a resource for people with chronic illnesses to support their independent self-management with rehabilitation strategies.

DETAILED DESCRIPTION:
Background: The global rise in chronic conditions and aging is associated with increased disability. Rehabilitation self-management (SM) strategies assist people with chronic conditions adjust to and manage their daily function. Technological interventions have the potential to increase the accessibility, availability and affordability of rehabilitation SM supports. IAMABLE is an evidence- and web-based app developed and tested by rehabilitation researchers. This app needs to be tested within a community context with consideration of implementation factors. Goals: The primary aim of this study is to assess the feasibility of conducting a fully powered RCT to assess the reach and effectiveness of the IAMABLE app in community-dwelling persons (45-76 years) with at least one musculoskeletal, cardiovascular or neurological chronic condition. The secondary aim is to assess adoption, implementation, and maintenance of the app in a population-based context.

Methods: We will conduct a hybrid (type 1) pilot effectiveness-implementation design guided by the REAIM framework. Assessments will be completed at baseline, 4- and 8-months. Participants (N=50) will be recruited in London, Hamilton, Kingston, Halifax and Winnipeg. Participants will be randomly allocated to receive the IAMABLE intervention (including access to modules, goal setting, self-assessments, tailored recommendations, and the "Ask a Therapist" feature) or a comparison group (with access to web-based general health information). For the effectiveness pilot, we will assess feasibility of conducting a fully-powered RCT. We will examine whether participants accessing the IAMABLE app for 4 months with a 4-month follow-up show greater improvement in self-reported function compared to persons in the comparison group. Secondary outcomes include quality of life, self-reported mobility, participation, efficacy with self-management, pain, fatigue, falls and health service use. To identify implementation, we will use integrated knowledge translation (quantitative and qualitative data from participants, therapists and app experts) engaged in expert panels using deliberative dialogue methods to evaluate adoption, use, and sustainability, and to formulate recommendations to improve implementation.

Research Team: Letts (NPA) and Richardson (PA) have collaborated for over 20 years in chronic disease SM research, incorporating technological innovations such as electronic self-monitoring, and web-based apps. Letts has expertise in community engagement and knowledge mobilization. Richardson has run numerous randomized trials. Co-applicants MacDermid and Colquhoun have expertise in implementation research. Co-applicants at each site will support participant recruitment and intervention delivery. All are rehabilitation researchers with expertise in chronic disease management; the team includes trainees, early career researchers and senior mentors. Patient partners will support recruitment and implementation research components. The team includes an expert in mobile app development and a statistician with expertise in pilot studies and trial methodology. Expected Outcomes: This research will demonstrate feasibility to determine if IAMABLE improves function and well-being of people with chronic conditions. Recommendations emerging from the study will support optimization of implementation of the app. Results will inform a fully powered trial embedded within a hybrid type 2 effectiveness implementation trial.

ELIGIBILITY:
Inclusion Criteria:

* is community-dwelling, has access to a computer or mobile device, has an email address, is able to follow directions in English, self-reports at least one of three types of prevalent chronic conditions associated with disability that frequently require rehabilitation supports (i.e., musculoskeletal, cardiovascular, and neurological conditions), responds "somewhat easily" or "very easily" to questions on the Modified Computer Proficiency Questionnaire (MCPQ-12).

Exclusion Criteria:

* scores < 11/15 on the Montreal Cognitive Assessment (MoCA) 5-Minute Test (Version 2.1).

Ages: 44 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-25 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility - Recruitment | Baseline
  Recruitment will be assessed by documenting the number of individuals who 1) express interest in participating, 2) were deemed eligible during telephone screening, 3) declined participation (and reasons for doing so), 4) were eligible at the baseline evaluation, and 5) withdrew consent after baseline assessment (and reasons of doing so). (Criterion: ≥75% of eligible participants recruited).
Feasibility - Response outcome adherence | Baseline
  Response outcome adherence will be measured by completion of secondary outcomes (Criterion: ≥80%).
Feasibility - Attrition | Baseline
  Attrition will be quantified throughout the study period as the number of participants who complete the outcome measures at the 3 timepoints (Criterion: ≤ 20% of participants enrolled withdrawn).
Feasibility - Program adherence | 4 months
  Program adherence will be quantified throughout the intervention period by documenting participant adherence to the protocol (e.g., # interactions with the app and frequency) (Criteria: at least one goal set, one module reviewed, two action plans completed).
Feasibility - Treatment fidelity | 4 months
  Treatment fidelity will be measured by monitoring therapists' responses when prompted by participants (Ask a Therapist feature) for timeliness of response being within 2 business days for any participant request (Criterion: ≥90% response within 2 days). We will audit 50% of the therapists' recommendations which will be de-identified (Criterion: ≥85% align with evidence-based modules and best evidence).
Feasibility - Adverse events | 4 months
  Adverse events and harms, including but not limited to muscle stiffness, soreness, injuries, or falls, will be documented throughout the intervention period. (Criterion: 0 serious adverse events related to module activities).
Feasibility - Response outcome adherence | 4 months
  Response outcome adherence will be measured by completion of secondary outcomes (Criterion: ≥80%).
Feasibility - Attrition | 4 months
  Attrition will be quantified throughout the study period as the number of participants who complete the outcome measures at the 3 timepoints (Criterion: ≤ 20% of participants enrolled withdrawn).
Feasibility - Response outcome adherence | 8 months
  Response outcome adherence will be measured by completion of secondary outcomes (Criterion: ≥80%).
Feasibility - Attrition | 8 months
  Attrition will be quantified throughout the study period as the number of participants who complete the outcome measures at the 3 timepoints (Criterion: ≤ 20% of participants enrolled withdrawn).

SECONDARY OUTCOMES:
Effectiveness - Self-reported physical function | Baseline
  Self-reported physical function will be measured using the Patient Specific Functional Scale (PSFS), an outcome measure used in patients with varying levels of independence.
Effectiveness - Patterns of mobility | Baseline
  Patterns of mobility will be evaluated using the Life-Space Assessment (LSA) Questionnaire, which assesses five space levels visited by the participant in the four weeks prior to the assessment.
Effectiveness - Participation | Baseline
  Participation will be assessed using the Computer Adaptive Testing (CAT) version of the Late Life Disability Instrument (LLDI-CAT). The LLDI measures limitations in perceived ability to perform social and instrumental roles.
Effectiveness - Knowledge, skill and confidence for SM | Baseline
  Knowledge, skill and confidence for SM will be measured using the Self-Efficacy for Managing Chronic Disease 6-item Scale (SES-6C), a measure of how confident patients with chronic disease are in managing fatigue, physical discomfort/pain, emotional distress, and activities needed to manage health conditions.
Effectiveness - Pain-related functional impairment | Baseline
  Pain-related functional impairment will be measured using the Brief Pain Inventory (BPI) Interference Scale. The BPI contains 7 domains, including general activity, mood, and walking ability.
Effectiveness - Fatigue | Baseline
  Fatigue will be assessed using the Checklist of Individual Strength (CIS), which assesses four dimensions of fatigue, fatigue severity, concentration problems, reduced motivation and activity.
Effectiveness - Quality of life | Baseline
  Quality of life will be measured using the SF-12, a widely used health profile in clinical trials with high test-retest reliability and responsiveness. Preference-based scores can be obtained from the SF-12, which can be used to calculate quality-adjusted life years (QALYs) for cost-utility analysis.
Effectiveness - Change in self-reported physical function | 4 months
  Self-reported physical function will be measured using the Patient Specific Functional Scale (PSFS), an outcome measure used in patients with varying levels of independence.
Effectiveness - Change in patterns of mobility | 4 months
  Patterns of mobility will be evaluated using the Life-Space Assessment (LSA) Questionnaire, which assesses five space levels visited by the participant in the four weeks prior to the assessment.
Effectiveness - Change in participation | 4 months
  Participation will be assessed using the Computer Adaptive Testing (CAT) version of the Late Life Disability Instrument (LLDI-CAT). The LLDI measures limitations in perceived ability to perform social and instrumental roles.
Effectiveness - Change in knowledge, skill and confidence for SM | 4 months
  Knowledge, skill and confidence for SM will be measured using the Self-Efficacy for Managing Chronic Disease 6-item Scale (SES-6C), a measure of how confident patients with chronic disease are in managing fatigue, physical discomfort/pain, emotional distress, and activities needed to manage health conditions.
Effectiveness - Change in pain-related functional impairment | 4 months
  Pain-related functional impairment will be measured using the Brief Pain Inventory (BPI) Interference Scale. The BPI contains 7 domains, including general activity, mood, and walking ability.
Effectiveness - Change in fatigue | 4 months
  Fatigue will be assessed using the Checklist of Individual Strength (CIS), which assesses four dimensions of fatigue, fatigue severity, concentration problems, reduced motivation and activity.
Effectiveness - Change in quality of life | 4 months
  Quality of life will be measured using the SF-12, a widely used health profile in clinical trials with high test-retest reliability and responsiveness. Preference-based scores can be obtained from the SF-12, which can be used to calculate quality-adjusted life years (QALYs) for cost-utility analysis.
Effectiveness - Healthcare utilization | 4 months
  Healthcare utilization data will be collected using a survey we have used in other clinical trials; this will contribute to planned cost-effectiveness.
Effectiveness - Change in self-reported physical function | 8 months
  Self-reported physical function will be measured using the Patient Specific Functional Scale (PSFS), an outcome measure used in patients with varying levels of independence.
Effectiveness - Change in patterns of mobility | 8 months
  Patterns of mobility will be evaluated using the Life-Space Assessment (LSA) Questionnaire, which assesses five space levels visited by the participant in the four weeks prior to the assessment.
Effectiveness - Change in participation | 8 months
  Participation will be assessed using the Computer Adaptive Testing (CAT) version of the Late Life Disability Instrument (LLDI-CAT). The LLDI measures limitations in perceived ability to perform social and instrumental roles.
Effectiveness - Change in knowledge, skill and confidence for SM | 8 months
  Knowledge, skill and confidence for SM will be measured using the Self-Efficacy for Managing Chronic Disease 6-item Scale (SES-6C), a measure of how confident patients with chronic disease are in managing fatigue, physical discomfort/pain, emotional distress, and activities needed to manage health conditions.
Effectiveness - Change in pain-related functional impairment | 8 months
  Pain-related functional impairment will be measured using the Brief Pain Inventory (BPI) Interference Scale. The BPI contains 7 domains, including general activity, mood, and walking ability.
Effectiveness - Change in fatigue | 8 months
  Fatigue will be assessed using the Checklist of Individual Strength (CIS), which assesses four dimensions of fatigue, fatigue severity, concentration problems, reduced motivation and activity.
Effectiveness - Change in quality of life | 8 months
  Quality of life will be measured using the SF-12, a widely used health profile in clinical trials with high test-retest reliability and responsiveness. Preference-based scores can be obtained from the SF-12, which can be used to calculate quality-adjusted life years (QALYs) for cost-utility analysis.
Effectiveness - Healthcare utilization | 8 months
  Healthcare utilization data will be collected using a survey we have used in other clinical trials; this will contribute to planned cost-effectiveness.

OTHER OUTCOMES:
Reach | 8 months
  Reach will be measured by the number of participants who are given access to initiate use of the app.
Adoption - Acceptability | 8 months
  Acceptability will be measured using the Service User Technology Acceptability Questionnaire. It has 22 items and 6 domains: perceived benefit, privacy and discomfort, care personnel concerns, app as a substitution, and satisfaction.
Adoption - Satisfaction | 8 months
  Satisfaction with the IAMABLE app will be measured using the 14-item mHealth Satisfaction Questionnaire.
Implementation | 8 months
  Study feasibility data on program adherence, treatment fidelity, and adverse events and harms will contribute to our understanding of implementation.
Sustainability | 8 months
  Individual interviews will be conducted at the end of 8 months to explore participants' experience of using the app over the intervention period. Data compiled re: adherence, acceptability, satisfaction and implementation will be compiled to support development of a sustainability plan for the IAMABLE app.

CONTACTS AND LOCATIONS:
Overall Officials: Lori Letts, PhD, Principal Investigator — McMaster University; Julie Richardson, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
All IPD related to publication results
Supporting Information: Study Protocol, SAP
Time Frame: IPD will be available at the time of publication and for 24 months.
Access Criteria: Qualified researchers engaging in independent scientific research.